CLINICAL TRIAL: NCT03958929
Title: A Randomized Controlled Trial on the Impact of an Educational Video on Satisfaction After Glaucoma Surgery in Urban and Rural China
Brief Title: Impact of an Educational Video on Satisfaction After Glaucoma Surgery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: change study sites
Sponsor: Sun Yat-sen University (Other)
Collaborators: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Congdon Nathan, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-074-K-73
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma
Keywords: glaucoma surgery; educational intervention; satisfaction; rural
MeSH Terms: conditions — Glaucoma; Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): Subjects will be asked to watch a 5-10 min education film two times (pre-op one day and post-op one day).
  Interventions: Other: Educational Video
- Control group (No Intervention): Standard patient procedure that includes a pre-operative discussion with an ophthalmologist about glaucoma surgery, during which the surgeon gains the patient's informed consent. Subjects will not be asked to watch education film..

INTERVENTIONS:
Other: Educational Video — The film follows the journey of an elderly patient scheduled to undergo glaucoma surgery, beginning with a face-to-face Q&A health session with an eye doctor. After surgery, the patient talks about his post-operative eyesight and discusses the benefits of early diagnosis and glaucoma surgery for treatment with his community.
  Arms: Education group

SUMMARY:
Overall Objective: This study will assess whether an educational video is effective in increasing patient satisfaction with glaucoma surgery.

1. Investigate the impact of educational interventions on glaucoma patients' surgical satisfaction.
2. Investigate the post-operative satisfaction of rural glaucoma patients in county hospitals
3. Investigate the difference in postoperative satisfaction between urban and rural glaucoma patients in urban hospitals
4. Investigate other factors that influence postoperative glaucoma satisfaction.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness in China, as elsewhere in the world. In Chinese rural settings, where topical glaucoma medication is unlikely to be a practical and sustainable option, surgery is the primary treatment modality for glaucoma.

However, it is known that vision is quite likely to decline in the short to medium term after glaucoma surgery, and there are concerns that dis-satisfaction resulting from such vision changes might lead to negative social marketing, affecting uptake not only of glaucoma surgical care but other eye operations (principally cataract) as well. We propose to test the impact on post-operative satisfaction of a multi-media educational intervention designed to give patients a realistic expectation of their post operative course: glaucoma surgery is being performed NOT to improve vision, but do protect it from future harm, and vision may in fact decline for several weeks post operatively.

A randomized controlled design will be used, and subjects undergoing glaucoma surgery will be enrolled at 4 rural county hospitals in rural Guangdong province, and randomized to receive the intervention or usual care. The principal outcome will be subjective satisfaction on a previously-tested questionnaire instrument, administered pre-operatively and post-operatively on two occasions in the first month following surgery. Patients not returning post-operatively to the surgical facility will be contacted by telephone for administration of the questionnaire. Other facility- and patient-related clinical and personal factors expected to influence satisfaction will also be recorded, and adjusted for in all analyses.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years, glaucoma patients who do the peripheral iridectomy or trabeculotomy

Exclusion Criteria:

* patients who had been the trabeculotomy, vision≤0.05, severe psychotic disorders and dysgnosia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-10-10 (Estimated); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
The mean satisfaction outcome over two follow-up visits | 1 day, 1 week
  The primary outcome is the mean satisfaction score calculated by adding up the satisfaction scores at two follow-up visits: 1 day and 1 week after surgery and dividing the total by the number of scores. The satisfaction score will be assessed as a cumulative score.
  Composite outcome, in which multiple end points are combined, are frequently used as primary outcome measures in randomized trials and are often associated with increased statistical efficiency, although such measure may prove challenging for the interpretation of results. (Freemantle N, Calvert M, Wood J, Eastaugh J, Griffin C. Composite outcomes in randomized trials: greater precision but with greater uncertainty? JAMA. 2003; 289: 2554-2559)

SECONDARY OUTCOMES:
The rate of willingness to recommend surgery to a friend or relative with glaucoma | 1 day, 1 week
  The measurement method: questionnaire
Personality in both groups using Eysenck Personality Questionnaire-Revised Short Scale for Chinese (EPQ-RSC) access glaucoma patients personality | Baseline (before surgery)
  The measurement method: questionnaire. The questionnaire provides subscores for 5 categories (Short, Extraversion, Neuroticism, Psychoticism, Lie score), with a higher corresponding to a higher characterization of that particular trait.
Knowledge scores about glaucoma | Baseline (before surgery); 1 day and 1 week after surgery
  The measurement method: questionnaire.
  Mean knowledge scores is calculated by adding up the scores at two follow-up visits: 1 day and 1 week after surgery and dividing the total by the number of scores. Knowledge scores will be assessed as a cumulative score, and will be compared with the baseline pre-operative score.
Intraocular pressure in both groups | Baseline (before surgery); 1 day and 1 week after surgery
  Unit of Intraocular pressure is mmHg.
visual acuity in both groups | Baseline (before surgery); 1 day and 1 week after surgery
  Visual acuity testing use Snellen-based letter charts,such as a Snellen score of 6/12 (20/40), indicating an observer can resolve details as small 2 minutes of visual angle, corresponds to a LogMAR of 0.3 (since the base-10 logarithm of 2 is 0.3)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD,MPH, Principal Investigator — The Key Laboratory,Zhongshan Ophthalmic Center,Sun Yat-sen University; Yuanbo Liang, MD, PhD, Principal Investigator — The Eye Hospital, Wenzhou Medical University
Locations (1):
- Affiliated Eye Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03958929/Prot_SAP_000.pdf